CLINICAL TRIAL: NCT02785757
Title: The Challenge of Cancer-related Thromboembolic Disease: Can we Better Predict the Risk?
Brief Title: Cancer-related Thromboembolic Disease
Acronym: PROSPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012.788; 2013-A00065-40 (Other: ID-RCB)
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Adenocarcinoma
Keywords: adenocarcinoma; venous thromboembolism; thrombin generation assay
MeSH Terms: conditions — Adenocarcinoma; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with adenocarcinoma (Experimental): 60 Patients recently diagnosed with locally advanced or metastatic adenocarcinoma of any origin, who are scheduled for systemic chemotherapy
  Interventions: Other: Thrombin Generation Assay

INTERVENTIONS:
Other: Thrombin Generation Assay

SUMMARY:
Patients with cancer are at particularly high risk of venous thromboembolism (VTE). The guidelines therefore strongly recommend thromboprophylaxis but recent surveys clearly show that oncologists are reluctant to use it because of concern over bleeding, absence of validated risk stratification tools and uncertainties concerning the optimal thromboprophylaxis. Hence, it is a real challenge to identify the individual VTE risk of each cancer patient and individually tailor their thromboprophylaxis.

The study aims to identify thrombin generation test (TGT) as a reliable, standardized overall haemostasis assay that can be used to evaluate individual thrombosis risk

The secondary objectives are:

* To define the limits of TGT parameters that indicate thrombosis risk in cancer patients
* To evaluate values of other clotting activation markers in patients with cancer

Patients recently diagnosed with locally advanced or metastatic adenocarcinoma of any origin, who are scheduled for systemic chemotherapy, will be enrolled in the trial at baseline (Visit 1). Thrombin generating capacity will be measured within the first month following diagnosis and before the start of the chemotherapy (between Visit 1 and Visit 2) and subsequently at the end of the first cure line of chemotherapy (Visit 3). Patients will be followed up for a period of 1 year, or until the occurrence of a thromboembolic event. Two follow up visits are foreseen - 6-month (Visit 4) and 12-month (or at the end of trial - Visit 5) visits.

Patients eventually undergoing second-line chemotherapy during the course of the follow-up will remain on study.

The study will document all cases of symptomatic thromboembolic events together with the relevant diagnostic work-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes with locally advanced or metastatic adenocarcinoma of any origin, who are scheduled for systemic chemotherapy
* Subjects having signed Informed Consent prior to initiation of any study procedure
* Covered by a Health System

Exclusion Criteria:

* Known bleeding or thrombophilia disorders
* Eastern Cooperative Oncology Group (ECOG) performance status ≥ 3
* Patient immobilized
* Confirmed venous thromboembolism in the last 12 months
* Active bleeding or bleedings in the last 4 weeks requiring hospitalization, transfusion, or surgical intervention
* Anticoagulant therapy at the moment of first sampling (at least one day off for Heparines and DOAc; at least 5 days off for VKA is needed)
* Antiplatelet therapy at the moment of first sampling (only if PRP TGA can be performed at site)
* Severe hepatic insufficiency
* Life expectancy of less than 3 months
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-07-12 (Actual); Primary Completion 2024-02-12 (Estimated); Study Completion 2024-02-12 (Estimated)

PRIMARY OUTCOMES:
thrombin generation assay results | 7 months

SECONDARY OUTCOMES:
Clotting activation markers: thrombin-antithrombin complexes (TAT) | 7 months
Clotting activation markers: prothrombin fragment F1+2 | 7 months
Clotting activation markers: D-dimer | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Unité d'Hémostase Clinique Hôpital Louis Pradel, Bron, France